CLINICAL TRIAL: NCT04386915
Title: To Evaluate the Tolerability and Pharmacokinetics of GST-HG141 Tablets in Single-center, Randomized, Double-blind, Placebo-controlled Multiple-dose, Single-dose, Multiple-dose Phase Ia Clinical Trials in Healthy Subjects
Brief Title: Study on the Tolerance and Pharmacokinetics of GST-HG141 Tablets
Acronym: GST-HG141
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cosunter Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GST-2020-001
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Single-dose experimental group (Experimental): 50mg, 100mg, 200mg, 300mg, 400mg, 500mg need to complete a single-dose clinical study, each group of 10 subjects, of which 8 received test drugs, 2 received placebo. Each group was administered once, under the fasting condition of Day1, and the tolerance was evaluated on Day2 and Day4. Subjects in different dose groups were enrolled in turn, and the next set of trials was conducted on the premise that the previous set of tolerability assessments were tolerated. The actual completion of the final dose, depending on the test results.
  Interventions: Drug: GST-HG141 tablets
- Single-dose control group (Placebo Comparator): 50mg, 100mg, 200mg, 300mg, 400mg, 500mg need to complete a single-dose clinical study, each group of 10 subjects, of which 8 received test drugs, 2 received placebo.
  Interventions: Drug: Placebo
- Multi-dose experimental group (Experimental): According to the results of the single-dose study, it is planned to carry out multiple-dose studies in 1 to 3 dose groups at 100 mg, 200 mg, 300 mg, and 400 mg. A total of 12 subjects in each dose group, of which 10 received the test drug, 2 received placebo. It is necessary to decide the multiple administration method and dosage according to the result of single administration, which is initially determined to be once a day. After the first dose, Day3, Day6, and Day12 were evaluated for tolerance, and the next group of tests was conducted under the premise that the previous group of Day12 tolerance evaluation was tolerated.
  Interventions: Drug: GST-HG141 tablets
- Multi-dose control group (Placebo Comparator): According to the results of the single-dose study, it is planned to carry out multiple-dose studies in 1 to 3 dose groups at 100 mg, 200 mg, 300 mg, and 400 mg. A total of 12 subjects in each dose group, of which 10 received the test drug, 2 received placebo.
  Interventions: Drug: Placebo
- Food Impact Study Group A (Experimental): Group A was administered under the fasting condition of Day1 in the first cycle, and under the postprandial conditions of Day8 ~ Day15 in the second cycle. Group B was administered under the postprandial conditions of Day1 in the first cycle, and under the sky-abdominal conditions of Day8 ~ Day15 in the second cycle. The two cycles are cross-administered, and the cleaning period is 7 to 14 days. In group A, the tolerance evaluation was conducted on Day 2 and Day 4 after the first administration. After the first dose of group A is completed and the tolerability evaluation result is considered tolerable, the second cycle of this group and the first cycle of group B can be carried out.
  Interventions: Drug: GST-HG141 tablets
- Food Impact Study Group B (Experimental): Group A was administered under the fasting condition of Day1 in the first cycle, and under the postprandial conditions of Day8 ~ Day15 in the second cycle. Group B was administered under the postprandial conditions of Day1 in the first cycle, and under the sky-abdominal conditions of Day8 ~ Day15 in the second cycle. The two cycles are cross-administered, and the cleaning period is 7 to 14 days. In group A, the tolerance evaluation was conducted on Day 2 and Day 4 after the first administration. After the first dose of group A is completed and the tolerability evaluation result is considered tolerable, the second cycle of this group and the first cycle of group B can be carried out.
  Interventions: Drug: GST-HG141 tablets

INTERVENTIONS:
Drug: GST-HG141 tablets — This trial includes single-dose studies and multiple-dose studies, The single-dose study included six dose groups of 50 mg, 100 mg, 200 mg, 300 mg, 400 mg, and 500 mg. Based on the results of a single dose, select 1 to 3 doses from 100mg, 200mg, 300mg, and 400mg to conduct multiple dose studies.
  Arms: Food Impact Study Group A; Food Impact Study Group B; Multi-dose experimental group; Single-dose experimental group
Drug: Placebo — This trial includes single-dose studies and multiple-dose studies, The single-dose study included six dose groups of 50 mg, 100 mg, 200 mg, 300 mg, 400 mg, and 500 mg. Based on the results of a single dose, select 1 to 3 doses from 100mg, 200mg, 300mg, and 400mg to conduct multiple dose studies.
  Arms: Multi-dose control group; Single-dose control group

SUMMARY:
To Evaluate the Tolerability and Pharmacokinetics of GST-HG141 Tablets in Single-center, Randomized, Double-blind, Placebo-controlled Multiple-dose, Single-dose, Multiple-dose Phase Ia Clinical Trials in Healthy Subjects .

DETAILED DESCRIPTION:
This trial includes single-dose studies and multiple-dose studies, The single-dose study included six dose groups of 50 mg, 100 mg, 200 mg, 300 mg, 400 mg, and 500 mg. Based on the results of a single dose, select 1 to 3 doses from 100mg, 200mg, 300mg, and 400mg to conduct multiple dose studies. To evaluate the tolerance of GST-HG141 tablets in healthy subjects in single and multiple administrations, pharmacokinetic characteristics, drug metabolism and transformation, and the effect of food on GST-HG141 pharmacokinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent before the trial and fully understand the content, process and possible adverse reactions of the trial;
2. Ability to complete research in accordance with test plan requirements;
3. Subjects (including partners) are willing to take effective pregnancy avoidance measures within 6 months after screening to the last study drug administration;
4. Male and female healthy subjects aged 18 to 55 years (including 18 and 55 years old);
5. Male subjects weigh no less than 50 kg, and female subjects weigh no less than 45 kg. Body mass index (BMI) = body weight (kg) / height 2 (m2), body mass index is in the range of 18 ~ 28 kg / m2 (including critical value);
6. Physical examination, normal or abnormal vital signs have no clinical significance.

Exclusion Criteria:

1. Those who smoked more than 5 cigarettes per day in the 3 months before the trial;
2. Allergies (multiple drugs and food allergies);
3. Have a history of drug abuse and / or alcoholism (drink 14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine);
4. Blood donation or massive blood loss (> 450 mL) within three months before screening;
5. Take any drug that changes the activity of liver enzymes 28 days before screening;
6. Took any prescription drugs, over-the-counter drugs, any vitamin products, or herbs within 14 days before screening;
7. Those who have taken special diets (including dragon fruit, mango, grapefruit, etc.) or have vigorous exercise or other factors affecting drug absorption, distribution, metabolism, excretion, etc. within 2 weeks before screening;
8. Combined with inhibitors or inducers of CYP3A4, such as itraconazole, ketoconazole, etc.;
9. Major changes in diet or exercise habits recently;
10. Have taken the study drug or participated in the drug clinical trial within three months before taking the study drug;
11. Have a history of dysphagia or any gastrointestinal disease that affects drug absorption;
12. Have any disease that increases the risk of bleeding, such as hemorrhoids, acute gastritis, or gastric and duodenal ulcers;
13. Subjects who cannot tolerate a standard meal (two boiled eggs, a piece of buttered bacon toast, a box of fried potato strips, a cup of full-fat milk) (this strip is only applicable to subjects participating in post-meal trials);
14. Abnormal ECG has clinical significance;
15. Female subjects were breastfeeding during the screening period or during the trial or were preparing for pregnancy recently or had a positive serum pregnancy result;
16. Clinical laboratory examinations are abnormal and clinically significant, or the following diseases (including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, Immune, mental or cardiovascular disease);
17. Positive screening for viral hepatitis (including hepatitis B and C), AIDS antigen / antibody, and Treponema pallidum antibody;
18. Acute disease or concomitant medication occurs from the screening stage to before study medication;
19. Ingested chocolate, any caffeinated or xanthine-rich food or drink 24 hours before taking the study drug;
20. Have taken any alcohol-containing product within 24 hours before taking the study drug;
21. People who have a positive urine drug screen or have a history of drug abuse or have used drugs within the past five years;
22. The investigator believes that there are other subjects who are not suitable for participating in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Peak Plasma Concentration (Cmax) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
T1/2 | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Cl/F | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis

SECONDARY OUTCOMES:
Ae(0~120h) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis
Fe(0~120h) | Measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 and 120hours in single-dosing. In the multiple dose group, measured on -0.5, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 12, 24hours on Day1, more details in protocol.
  Plasma samples were collected at different points for pharmacokinetic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Junqi Niu, PHD, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The first hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No